CLINICAL TRIAL: NCT05235022
Title: After Cancer in the Military: What Happens After Long-term Sick Leave
Acronym: APCAM-CLDM
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PPRC07; 2021-A02180-41 (Other: IDRCB)
Record Dates: First submitted 2022-01-25; First posted 2022-02-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Cancer
Keywords: Long-term sick leave
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — The participants included in the study will have to answer:
  1. a questionnaire created specifically for the study concerning the possible difficulties encountered during their return to work,
  2. the Multidimensional Fatigue Inventory (MFI), a questionnaire assessing fatigue through 5 dimensions (general fatigue, physical fatigue, mental fatigue, reduced activity and reduced motivation).
  These 2 questionnaires will be filled during a 30-minute face-to-face or phone interview.

SUMMARY:
In recent decades, early diagnosis and improved treatment have led to increased survival for most people with cancer. This improved survival has led to more attention being paid to the quality of life of these people, and to their reintegration into social and professional life. In France, 3.8 million people are treated or in remission from cancer in 2017. Among the 400,000 new patients diagnosed with cancer each year in France, 160,000 (40%) are in professional activity.

Cancer treatments induce after-effects that can be felt several months or even years after the diagnosis and have an impact on life. In a study of patients in remission from cancer at 12 months after diagnosis, 47 to 53% of patients had changed jobs or stopped working. In another Finnish study, 26% of patients had decreased physical ability and 19% had decreased mental ability to work five years after cancer diagnosis.

In France, studies that have evaluated the impact of cancer on employment and the factors associated with return to work after cancer are still rare: the VICAN study showed that among people in work at the time of diagnosis, 20% were no longer working five years later.

With an estimated annual incidence of approximately 400 new cancers per year, the military population is also affected by cancer. Professional reintegration after cancer is of particular concern to the military. The specificity and requirements of the military condition can indeed make this reintegration more difficult. Regular or even intense physical activity is indeed essential but can be difficult after undergoing anti-cancer treatments. Moreover, external operations and many activities are conditioned by the obtaining of medical skills, which are sometimes incompatible with the state of health of patients recently treated for a neoplastic pathology. The studies previously carried out concerning the professional future after cancer do not seem to us to be transposable to the military population. To our knowledge, no study has evaluated occupational reintegration in military personnel after cancer.

The aim of this study is to evaluate the difficulties encountered during the post-cancer professional reintegration of military personnel in terms of fatigue, aptitude and advancement, in order to anticipate them and possibly remedy them. The identification of these difficulties will eventually allow to anticipate them and possibly to remedy them via an adapted post-cancer professional reintegration pathway.

ELIGIBILITY:
Inclusion Criteria:

* French military personnel who were placed on long-term sick leave for the management of a tumor pathology between January 2015 and December 2020,
* French-speaking.

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of French military personnel who were placed on long-term sick leave for the management of a tumor pathology between January 2015 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Description of the difficulties reported by the patients during their return to work after cancer | Until the end of the study (12 months)
  The primary outcome measure is descriptive. The purpose is to highlight the difficulties most often mentioned by patients during the interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Sainte-Anne, Toulon, France

IPD SHARING:
Plan to Share IPD: Undecided